CLINICAL TRIAL: NCT07255404
Title: A Phase II, Multi-site, Randomized, Open-label, Trial of BNT327 in Combination With Chemotherapy in Patients With Metastatic Pancreatic Cancer
Brief Title: A Clinical Trial Testing the Safety of BNT327 (an Investigational Drug) and How Well it Works When Combined With Chemotherapy for People Who Have Not Been Treated Yet for Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Bristol-Myers Squibb (Industry); BioNTech (Shanghai) Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-09
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: PDAC; Bispecific antibody; Metastatic pancreatic cancer; Immunotherapy; Immunotherapy in combination with chemotherapy; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor(-A) (VEGF-A)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1: Pumitamig (dose level 1) + chemotherapy (Experimental): Participants will be administered pumitamig plus chemotherapy regimen.
  Interventions: Drug: Pumitamig; Drug: mFOLFIRINOX
- Arm 2: Pumitamig (dose level 2) + chemotherapy (Experimental): Participants will be administered pumitamig plus chemotherapy regimen.
  Interventions: Drug: Pumitamig; Drug: mFOLFIRINOX
- Arm 3: Pumitamig (dose level 2) + chemotherapy (Experimental): Participants will be administered pumitamig plus chemotherapy regimen.
  Interventions: Drug: Pumitamig; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm 4A (exploratory): Pumitamig (dose level 2) + treatment of physician's choice chemotherapy (Experimental): Participants will be administered pumitamig plus chemotherapy regimen.
  Interventions: Drug: Pumitamig; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm 4B (exploratory): Pumitamig (dose level 2) + treatment of physician's choice chemotherapy (Experimental): Participants will be administered pumitamig plus chemotherapy regimen
  Interventions: Drug: Pumitamig; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Pumitamig — Intravenous (IV) infusion
  Other Names: BNT327; PM8002; BMS-986545
Drug: Nab-paclitaxel — IV infusion
  Arms: Arm 3: Pumitamig (dose level 2) + chemotherapy; Arm 4A (exploratory): Pumitamig (dose level 2) + treatment of physician's choice chemotherapy
Drug: Gemcitabine — IV infusion
  Arms: Arm 3: Pumitamig (dose level 2) + chemotherapy; Arm 4A (exploratory): Pumitamig (dose level 2) + treatment of physician's choice chemotherapy
Drug: mFOLFIRINOX — IV infusion
  Arms: Arm 1: Pumitamig (dose level 1) + chemotherapy; Arm 2: Pumitamig (dose level 2) + chemotherapy; Arm 4B (exploratory): Pumitamig (dose level 2) + treatment of physician's choice chemotherapy

SUMMARY:
This study will enroll adults with confirmed metastatic pancreatic ductal adenocarcinoma (PDAC, systemic PDAC treatment naïve), Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1, and adequate organ function. Participants will receive pumitamig (BNT327) in combination with chemotherapy.

DETAILED DESCRIPTION:
Participants will be assigned to treatment arms with modified (m) FOLFIRINOX administration (Treatment Arms 1 and 2) or the treatment arm with nab-paclitaxel + gemcitabine administration (Treatment Arm 3) based on the physician's choice of chemotherapy. Study participants assigned to arms with mFOLFIRINOX administration, will be randomized 1:1 to one of the two arms (Treatment Arms 1 or 2). Once enrollment of Treatment Arms 1 to 3 has been completed, enrollment into the exploratory cohorts (Treatment Arms 4A and 4B) will be opened.

There will be a screening period of up to 28 days, followed by a treatment period lasting up to 2 years. After administration of the last dose of study treatment, participants will be followed-up for safety for up to 90 days or until the participant initiates new anticancer treatment (e.g., systemic, radiotherapy/surgery). Thereafter, survival follow-up will be conducted until the participant dies or withdraws consent for survival status follow-up, loss of contact, or study termination (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed metastatic PDAC. A tissue sample, archival or fresh, must be provided during the screening period. In case it is not feasible to meet the required tumor tissue criteria, approval by the sponsor's medical monitor is needed for enrollment.
* Have not received prior systemic therapy for unresectable metastatic PDAC. For participants who have received prior induction chemotherapy, concurrent chemoradiotherapy, or adjuvant/neoadjuvant chemotherapy for curative-intent, the interval should be at least 6 months from the end of the last treatment to relapse.
* Have at least one measurable lesion as the targeted lesion based on RECIST v1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures) are not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system [CNS] metastasis should not be considered as a measurable lesion).
* Agree to discontinue strong inhibitors or inducers of cytochrome P450 enzyme (CYP3A), CYP2C8, glucuronosyltransferase 1 family, polypeptide A cluster 1A (UGT1A1) at least 2 weeks prior to starting study treatment, and change to other treatment regimens at screening if such drugs are used.

Exclusion Criteria:

* Have received any of the following therapies or drugs before study enrollment:

  * Have received prior systemic anticancer therapy for unresectable metastasis disease.
  * Any anticancer therapy, including systemic, palliative, biologic, immunostimulatory, or immunosuppressive treatment within 4 weeks (or five half-lives, whichever is longer) before starting study treatment.
  * PD(L)-1/VEGF bispecific antibody, including monotherapy with either category or combinations thereof.
  * Systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 14 days before starting study treatment. Exception: Excluding local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergies) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens).
  * Vaccinations with live attenuated vaccine(s) within 4 weeks before starting study treatment.
  * Broad-spectrum intravenous antibiotics therapy within 2 weeks before starting study treatment.
  * Any non-study investigational medicinal product within five half-lives of the first dose or within 4 weeks, whichever is longer, before initiation of study treatment in this study or ongoing participation in the active treatment phase of another interventional clinical study.
  * Antiplatelet drugs, such as aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine or cilostazol, etc., within 10 days before starting study treatment to avoid inclusion of participants who have used platelet aggregation inhibitors before the study.
* Have undergone major organ surgery (core needle biopsies are allowed >7 days before starting study treatment), open biopsy, significant trauma, or invasive dental procedures (such as dental implants) within 28 days before starting study treatment, or a planned/anticipated need for major surgery during the study treatment period. Placement of vascular infusion devices is allowed. Note: If participant has had major surgery, they must have recovered adequately from the toxicity and/or complications from the treatment before starting study treatment.
* Have received allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Have spinal cord compression or CNS metastases that are untreated and symptomatic or require treatment with corticosteroids or anticonvulsants for associated-symptom control. Exception: Treated brain metastases which are no longer symptomatic and for which no corticosteroid or anticonvulsant treatment is needed (the participant must have recovered from the acute toxic effect of radiotherapy).
* Have active autoimmune disease or history of autoimmune diseases with anticipated relapse (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for those with clinically stable autoimmune thyroid disease or type 1 diabetes mellitus.
* Have had other malignant tumors within 5 years before starting study treatment. Exception: Those who have been cured with local treatment (such as basal cell or squamous-cell carcinoma of the skin, superficial or noninvasive bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary carcinoma of thyroid and early-stage prostate cancer).
* Have heart conditions as specified in the protocol within 6 months before starting study treatment.
* Have uncontrolled hypertension or poorly controlled diabetic conditions as specified in the protocol before starting study treatment.
* History of myocardial infarction, unstable angina, arterial thrombosis or cerebrovascular accident within 6 months before starting study treatment.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism within 3 months prior to randomization, unless the participant has been fully treated (e.g., inferior vena cava filter placed) and/or adequately anticoagulated on a prophylactic dose.
* Have serious or non-healing wounds, ulcers, or (incompletely healed) bone fractures. This includes history (within 6 months before starting the study treatment) or risk of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess or esophageal and gastric varices, or acute gastrointestinal bleeding. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Have significant risk of hemorrhage (in the opinion of the investigator) or evidence of major coagulation disorders as specified in the protocol.
* Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Those with indwelling catheters (e.g., PleurX) are allowed.
* Participants with a history of serious Grade 3 or higher immune-related adverse events (irAEs) that led to treatment discontinuation of a prior immunotherapy. Participants with a history of Grade 3 or higher irAEs that did not lead to treatment discontinuation of a prior immunotherapy may be enrolled at the investigator's discretion.
* Have adverse events (AEs) from prior antitumor therapy that have not returned to Grade 1 (graded by CTCAE v5.0 criteria) or below (unless the investigator determines that certain AEs pose no safety risk to participants, such as hair loss, Grade 2 peripheral neuropathy or stable hypothyroidism under hormone replacement therapy).
* Have gastrointestinal symptoms or conditions as specified in the protocol.
* History of serious allergic diseases, history of serious allergy to drugs (including unlisted investigational drug) or known allergy or intolerance to any ingredient of the study treatment.
* Have superior vena cava syndrome or symptoms of spinal cord compression.
* Have active, or a history of, pneumonitis requiring treatment with steroids, or have active or a history of interstitial lung disease. Those with a history of pulmonary fibrosis or with currently diagnosed severe lung diseases such as interstitial pneumonia, pneumoconiosis, chemical pneumonitis, or any other condition resulting in significant impairment in lung function. Exception: Asymptomatic interstitial changes caused by previous radiotherapy, chemotherapy, or other factors such as smoking are allowed.
* Have a known history of tuberculosis that was not successfully treated.
* Have active syphilis. Participants with inactive previous infection could be eligible: Infection with a positive non-specific antibody test for syphilis (e.g., TRUST [Toluidine Red Unheated Serum Test], Rapid Plasma Reagin [RPR], TP-PA [Treponema pallidum Particle Agglutination]) or have a positive syphilis-specific antibody test (e.g., TPPA) (a positive "syphilis-specific antibody test" but a negative "non-specific antibody test for syphilis" for more than 1 year) infection.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall response rate | Up to 24 months
  For each treatment arm. Defined as the percentage of study participants in whom a confirmed complete response (CR) or confirmed partial response (PR) (assessed by the investigator per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) is observed as best overall response.
Occurrence of treatment emergent adverse events (TEAEs) by severity | From the first dose of study treatment until 90 days after the last dose of study treatment (up to 32 months).
  According to (US National Cancer Institute) Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v5.0]). By relationship and for each treatment arm.
Occurrence of dose interruptions, reductions, and discontinuations due to TEAEs | Up to 24 months after first dose
  For each treatment arm.

SECONDARY OUTCOMES:
Disease control rate | Up to 24 months
  Defined as the percentage of study participants in whom a confirmed CR or confirmed PR or stable disease (SD), (per RECIST v1.1, SD assessed at least 6 weeks after randomization/assignment to treatment) is observed as best overall response.
Duration of response | Up to 30 months
  Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (disease progression as assessed by the investigator per RECIST v1.1), or death from any cause, whichever occurs first.
Progression free survival | Up to 32 months
  Defined as the time from randomization/assignment to treatment to first documented tumor progression (disease progression assessed by investigator per RECIST v1.1), or death from any cause, whichever occurs first.
Overall survival | Up to 32 months
  Defined as the time from participant randomization/assignment to treatment to death from any cause.
Pharmacokinetic (PK) assessment: Maximum concentration (Cmax) derived from serum concentration of pumitamig | Up to 6 months from first dose of study treatment
  At Cycle 1 and Cycle 6 as data permits.
PK assessment: Minimum concentration (Cmin) derived from serum concentration of pumitamig | Up to 6 months from first dose of study treatment
  At Cycle 1 and Cycle 6 as data permits.
Incidence of detectable pumitamig anti-drug antibodies in serum | Up to 32 months
  From before the first dose of study treatment until the last survival follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No